CLINICAL TRIAL: NCT00765674
Title: An 8 Week, Double-blind, Randomized, Parallel Group, Active-controlled Study to Evaluate the Efficacy and Safety of the Combination of Aliskiren/Amlodipine/Hydrochlorothiazide in Patients With Moderate to Severe Hypertension
Brief Title: Efficacy and Safety of Aliskiren/Amlodipine/Hydrochlorothiazide in Patients With Moderate-severe Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSAH100A2302
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Results first posted 2011-05-09 (Estimated); Last update posted 2011-05-09 (Estimated); Status verified 2011-04

CONDITIONS: Hypertension
Keywords: aliskiren; antihypertensive; hypertension; renin inhibitor; moderate-severe hypertension
MeSH Terms: conditions — Hypertension | interventions — aliskiren; Amlodipine; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Aliskiren / amlodipine (Experimental): Patients received an aliskiren 150 mg tablet plus an amlodipine 5 mg capsule for 4 weeks and then were force titrated up to aliskiren 300 mg plus amlodipine 10 mg for the remaining 4 weeks of the study. During the 8 weeks, patients also received a placebo tablet and a placebo capsule. Patients took a total of 4 pills each day orally with water in the morning at approximately 8:00 am, except on the morning of a study visit when they took their study medications after all visit procedures and assessments had been completed.
  Interventions: Drug: Aliskiren; Drug: Amlodipine; Drug: Placebo
- Aliskiren / hydrochlorothiazide (Experimental): Patients received an aliskiren 150 mg tablet plus a hydrochlorothiazide 12.5 mg capsule for 4 weeks and then were force titrated up to aliskiren 300 mg plus hydrochlorothiazide 25 mg for the remaining 4 weeks of the study. During the 8 weeks, patients also received a placebo capsule and a placebo tablet. Patients took a total of 4 pills each day orally with water in the morning at approximately 8:00 am, except on the morning of a study visit when they took their study medications after all visit procedures and assessments had been completed.
  Interventions: Drug: Aliskiren; Drug: Hydrochlorothiazide (HCTZ); Drug: Placebo
- Amlodipine / hydrochlorothiazide (Experimental): Patients received an amlodipine 5 mg capsule plus a hydrochlorothiazide 12.5 mg capsule for 4 weeks and then were force titrated up to amlodipine 10 mg plus hydrochlorothiazide 25 mg for the remaining 4 weeks of the study. During the 8 weeks, patients also received 2 placebo tablets. Patients took a total of 4 pills each day orally with water in the morning at approximately 8:00 am, except on the morning of a study visit when they took their study medications after all visit procedures and assessments had been completed.
  Interventions: Drug: Amlodipine; Drug: Hydrochlorothiazide (HCTZ); Drug: Placebo
- Aliskiren / amlodipine / hydrochlorothiazide (Experimental): Patients received an aliskiren 150 mg tablet, a HCTZ 12.5 mg capsule and a placebo capsule for the first 3 days of treatment. Amlodipine 5 mg was then added for the remainder of the first 4 weeks of treatment. At the end of 4 weeks, patients were force titrated up to aliskiren / amlodipine / hydrochlorothiazide 300/10/25 mg for the remaining 4 weeks of the study. During the 8 weeks, patients also received a placebo tablet. Patients took a total of 4 pills each day orally with water in the morning at approximately 8:00 am, except on the morning of a study visit when they took their study medications after all visit procedures and assessments had been completed.
  Interventions: Drug: Aliskiren; Drug: Amlodipine; Drug: Hydrochlorothiazide (HCTZ); Drug: Placebo

INTERVENTIONS:
Drug: Aliskiren — 150 and 300 mg tablets
  Arms: Aliskiren / amlodipine; Aliskiren / amlodipine / hydrochlorothiazide; Aliskiren / hydrochlorothiazide
Drug: Amlodipine — 5 and 10 mg capsules
  Arms: Aliskiren / amlodipine; Aliskiren / amlodipine / hydrochlorothiazide; Amlodipine / hydrochlorothiazide
Drug: Hydrochlorothiazide (HCTZ) — 12.5 and 25 mg capsules
  Arms: Aliskiren / amlodipine / hydrochlorothiazide; Aliskiren / hydrochlorothiazide; Amlodipine / hydrochlorothiazide
Drug: Placebo — tablet
Drug: Placebo — capsules
  Arms: Aliskiren / amlodipine; Aliskiren / hydrochlorothiazide

SUMMARY:
This study evaluated the efficacy (blood pressure lowering effect) and safety of aliskiren/amlodipine/hydrochlorothiazide in patients with moderate to severe hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18 years of age or older
* msDBP and msSBP requirements:

  * 3A:

    * Diagnosis of moderate to severe hypertension (msSBP ≥ 160 mmHg and < 200 mmHg, and/or msDBP ≥ 100 mmHg and < 120 mmHg) at Visits 4, 5 or 6 (Qualifying BP visit)
    * In addition, at the visit immediately prior to the above qualifying visit, patients were also to have msSBP ≥ 145 mmHg and < 200 mmHg and msDBP ≥ 95 mmHg and < 120 mmHg) at Visits 3, 5 or 5.
    * Patients had to meet the above two sets of requirements at subsequent adjacent visits, i.e. either Visits 3 and 4, Visits 4 and 5, or Visits 5 and 6.
  * OR
  * 3B:

    * msSBP ≥ 180 mmHg and < 200 mmHg with msDBP ≥ 95 mmHg and < 120 mmHg, or msDBP ≥ 110 mmHg and < 120 mmHg with msSBP ≥ 150 mmHg and < 200 mmHg after at least one week of treatment with placebo (Visit 3 and on).

Exclusion Criteria:

* Continued use of anti-hypertensive medicines or use of 4 or more hypertensive medicines at study start
* Patients with an msSBP ≥ 200 mmHg or msDBP ≥ 120 mmHg at any time during the placebo run-in period were to be discontinued from the study.
* Extremely elevated (defined) blood pressure at any point during the study
* Pregnant or lactating women
* Pre-menopausal women not taking accepted form of birth control
* History or evidence of secondary form of hypertension
* History of cardiovascular conditions

Other protocol-defined inclusion/exclusion criteria applied to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1191 (Actual)
Dates: Start 2008-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- Investigative Site, Denver, Colorado, United States
- Investigative Site, Sydney, Australia
- Investigative Site, Ottawa, Canada
- Investigative Site, Copenhagen, Denmark
- Investigative Site, Berlin, Germany
- Investigative Site, Jerusalem, Israel
- Investigative Site, Rome, Italy
- Investigative Site, Riga, Latvia
- Investigative Site, Vilnius, Lithuania
- Investigative Site, Bucharest, Romania
- Investigative Site, Stockholm, Sweden
- Investigative Site, Ankara, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the single-blind period, 1909 patients were enrolled, 1189 completed, and 720 discontinued. Of the 1191 randomized patients, 2 patients were randomized by error and discontinued in the single-blind period without taking double-blind medication.
Period: Overall Study
Arm/Group | Aliskiren / Amlodipine | Aliskiren / Hydrochlorothiazide | Amlodipine / Hydrochlorothiazide | Aliskiren / Amlodipine / Hydrochlorothiazide
Started | 287 | 298 (1 patient was randomized in error and discontinued without taking any double-blind study medication.) | 296 | 310 (1 patient was randomized in error and discontinued without taking any double-blind study medication.)
Completed | 266 | 276 | 279 | 285
Not Completed | 21 | 22 | 17 | 25
Not completed — Adverse Event | 7 | 2 | 8 | 11
Not completed — Abnormal Laboratory Value(s) | 0 | 0 | 1 | 0
Not completed — Abnormal Test Procedure Result(s) | 1 | 3 | 1 | 2
Not completed — Lack of Efficacy | 2 | 3 | 1 | 2
Not completed — Protocol Violation | 2 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 7 | 3 | 8
Not completed — Lost to Follow-up | 4 | 6 | 2 | 1
Not completed — Randomized in Error - No Study Drug | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren / Amlodipine | Aliskiren / Hydrochlorothiazide | Amlodipine / Hydrochlorothiazide | Aliskiren / Amlodipine / Hydrochlorothiazide | Total
Number analyzed (Participants) | 287 | 298 | 296 | 310 | 1191
Age Continuous [Mean (Standard Deviation); unit: years] | 54.4 (11.33) | 55.5 (10.75) | 55.1 (10.86) | 55.4 (10.54) | 55.1 (10.86)
Age, Customized [Number; unit: participants]
  < 65 years | 237 | 242 | 233 | 251 | 963
  >=65 years | 50 | 56 | 63 | 59 | 228
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 123 | 110 | 123 | 471
  Male | 172 | 175 | 186 | 187 | 720

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Sitting Systolic Blood Pressure (msSBP) From Baseline to End of Study (Week 8)
Description: Blood pressure (BP) was measured at trough (24±3 hours post-dose). The arm in which the highest sitting diastolic BP was found at study entry was used for all subsequent readings. If there was < 0.5 mmHg difference in BP between the 2 arms, the non-dominant arm was used. At each visit, after the patient was in a sitting position with the back supported and both feet placed on the floor for 5 minutes, systolic and diastolic BP were measured 3 times with an automated BP monitor and appropriate size cuff. Means of the 3 measurements were calculated. A negative change indicates lowered BP.
Time Frame: Baseline to end of study (Week 8)
Population: Full analysis set population: All randomized patients who had post-baseline efficacy measurements.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren / Amlodipine | Aliskiren / Hydrochlorothiazide | Amlodipine / Hydrochlorothiazide | Aliskiren / Amlodipine / Hydrochlorothiazide
Number analyzed (Participants) | 282 | 296 | 295 | 308
mmHg | -31.37 (0.90) | -27.99 (0.88) | -30.77 (0.88) | -37.92 (0.86)

2. Secondary Outcome: Change in Mean Sitting Diastolic Blood Pressure (msDBP) From Baseline to End of Study (Week 8)
Description: as for outcome 1
Time Frame: Baseline to end of study (Week 8)
Population: Full analysis set population: All randomized patients who had post-baseline efficacy measurements.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren / Amlodipine | Aliskiren / Hydrochlorothiazide | Amlodipine / Hydrochlorothiazide | Aliskiren / Amlodipine / Hydrochlorothiazide
Number analyzed (Participants) | 282 | 296 | 295 | 308
mmHg | -18.03 (0.57) | -14.32 (0.55) | -17.03 (0.55) | -20.63 (0.54)

3. Secondary Outcome: Percentage of Patients Achieving Blood Pressure Control at the End of the Study (Week 8)
Description: Blood pressure control was defined as a msSBP/msDBP < 140/90 mmHg at the end of the study (Week 8). Blood pressure (BP) was measured at trough (24±3 hours post-dose). The arm in which the highest sitting diastolic BP was found at study entry was used for all subsequent readings. At each visit, after the patient was in a sitting position with the back supported and both feet placed on the floor for 5 minutes, systolic and diastolic BP were measured 3 times with an automated BP monitor and appropriate size cuff. Means of the 3 measurements were calculated.
Time Frame: End of study (Week 8)
Population: Full analysis set population: All randomized patients who had post-baseline efficacy measurements.
Measure: Number; unit: Percentage of patients
Arm/Group | Aliskiren / Amlodipine | Aliskiren / Hydrochlorothiazide | Amlodipine / Hydrochlorothiazide | Aliskiren / Amlodipine / Hydrochlorothiazide
Number analyzed (Participants) | 283 | 296 | 295 | 192
Percentage of patients | 41.3 | 33.1 | 39.0 | 62.3

4. Secondary Outcome: Change in Mean 24-hour Ambulatory Systolic and Diastolic Blood Pressure From Baseline to End of Study (Week 8)
Description: Twenty-four hour ambulatory blood pressure monitoring (ABPM) was performed in a subset of patients twice during the study, once at baseline and again at Week 8. The ABPM device was placed on the non-dominant arm between 7:00 and 10:00 am and verification readings obtained. If they were successful, the investigator initiated the 24 hour reading and instructed the patient regarding ABPM procedures. On the next day, the ABPM device was removed if it had been worn for a minimum of 24 hours. The ABPM data were downloaded and evaluated on site.
Time Frame: Baseline to end of study (Week 8)
Population: Full analysis set population: All randomized patients who had post-baseline efficacy measurements.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren / Amlodipine | Aliskiren / Hydrochlorothiazide | Amlodipine / Hydrochlorothiazide | Aliskiren / Amlodipine / Hydrochlorothiazide
Number analyzed (Participants) | 138 | 155 | 136 | 147
mmHg
  Systolic BP | -20.30 (0.52) | -16.27 (0.51) | -18.67 (0.53) | -25.29 (0.51)
  Diastolic BP | -13.29 (0.36) | -9.57 (0.35) | -11.20 (0.37) | -15.90 (0.35)

ADVERSE EVENTS:
Time Frame: During the 8 week double blind treatment
Description: Safety Set. All patients who received double-blind trial medication.
Arm/Group | Aliskiren / Amlodipine | Aliskiren / Hydrochlorothiazide | Amlodipine / Hydrochlorothiazide | Aliskiren / Amlodipine / Hydrochlorothiazide
Serious Adverse Events (participants affected / at risk) | 3/287 | 2/297 | 2/295 | 6/309
Other Adverse Events (participants affected / at risk) | 32/287 | 17/297 | 26/295 | 29/309
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren / Amlodipine (N=287) | Aliskiren / Hydrochlorothiazide (N=297) | Amlodipine / Hydrochlorothiazide (N=295) | Aliskiren / Amlodipine / Hydrochlorothiazide (N=309)
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 1
Arrhythmia supraventricular (Cardiac disorders) | 0 | 0 | 0 | 1
Goitre (Endocrine disorders) | 0 | 0 | 0 | 1
Hepatitis A (Infections and infestations) | 1 | 0 | 0 | 0
Tubo-ovarian abscess (Infections and infestations) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Psychosomatic disease (Psychiatric disorders) | 0 | 0 | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren / Amlodipine (N=287) | Aliskiren / Hydrochlorothiazide (N=297) | Amlodipine / Hydrochlorothiazide (N=295) | Aliskiren / Amlodipine / Hydrochlorothiazide (N=309)
Oedema peripheral (General disorders) | 23 | 6 | 12 | 22
Headache (Nervous system disorders) | 9 | 12 | 15 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.